CLINICAL TRIAL: NCT01283009
Title: CSP #574 - Evaluate the Safety and Efficacy of Methylprednisolone in Hospitalized Veterans With Severe Community-Acquired Pneumonia
Brief Title: Extended Steroid in Use in Community Acquired Pneumonia (CAP)(e)
Acronym: ESCAPe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 574
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Community Acquired Respiratory Disease Syndrome
Keywords: pneumoniae
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Inactive substance (Placebo Comparator): Inactive substance
  Interventions: Drug: Inactive Substance
- Arm 2: Methylprednisolone (Active Comparator): Methylprednisolone
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Inactive Substance — Inactive Substance will be given in a double-blind fashion for 20 full days. The treatment course includes a bolus dose on the day of randomization, 7 days of full dose (40 mg/day), 7 days of half dose (20 mg/day), and 6 days of tapering doses (12 mg/day and 4 mg/day).
  Arms: Arm 1: Inactive substance
Drug: Methylprednisolone — Methylprednisolone will be given in a double-blind fashion for 20 full days. The treatment course includes a bolus dose on the day of randomization, 7 days of full dose (40 mg/day), 7 days of half dose (20 mg/day), and 6 days of tapering doses (12 mg/day and 4 mg/day).
  Other Names: Medrol
  Arms: Arm 2: Methylprednisolone

SUMMARY:
The goal of the study is to determine whether providing early treatment with a glucocorticoid drug, called methylprednisolone, will improve survival in critically ill patients with severe community-acquired pneumonia (CAP). Pneumonia develops when bacteria and other agents invade the lungs. The body's immune system creates a response to produce inflammation to kill the bacteria. A moderate amount of inflammation is beneficial. But, in patients sick enough to be admitted to the ICU, inflammation is frequently out of control. When the body cannot regulate inflammation vital organs (brain, heart, lung, kidney, liver) may be damaged, contributing to death or residual organ damage for those who survive. Glucocorticoids help reduce inflammation. Recent studies have shown that when the body is unable to produce sufficient amounts of glucocorticoids, inflammation can get out of control. Under these circumstances, glucocorticoids given in small doses may help aid the body's ability to reduce inflammation and improve recovery. In a small preliminary trial, glucocorticoid treatment, in addition to standard antibiotic treatment, sped up recovery from pneumonia. It also decreased the length of hospital stay, and increased survival. This Cooperative Studies Program (CSP) study will be the first large-scale, prospective, randomized clinical trial evaluating whether or not this treatment improves recovery.

In this study, at each site, patients with severe CAP will be assigned to one of two treatment groups. One group will receive methylprednisolone and the other will receive a placebo (an inert substance that will look like the drug). The investigators have chosen a total duration of treatment of 20 days (7 days full dose followed by slow reduction over 13 days) to prevent relapse of inflammation and allow the body to recover its own ability to produce glucocorticoid. All patients will also receive standardized management of CAP in accordance with current practice guidelines. The study will take into consideration when assigning the treatment each participating site, and whether or not the patient requires mechanical ventilation at the time of assignment. Patients will be followed clinically for 180 days. The primary outcome is all cause 60-day mortality. Secondary outcomes are (1) in-hospital morbidity-mortality, including ventilator-free days, multiorgan dysfunction syndrome (MODS)-free days, duration of ICU and hospital stay, and hospital discharge; and (2) posthospital discharge morbidity-mortality, including cardiovascular complications, functional and general health status in the first 180 days, rehospitalization, and mortality at 1 year. Serial blood samples will also be collected and stored for future translational research relating longitudinal inflammation markers to clinical outcomes.

This study will advance knowledge on the relationship between inflammation and long-term outcome in severe CAP.

DETAILED DESCRIPTION:
VA Cooperative Study #574 is designed to prospectively evaluate the efficacy of prolonged glucocorticoid (methylprednisolone) treatment on short- (in hospital) and long-term (after hospital discharge), morbidity and mortality in Veteran patients admitted to the Intensive Care Unit (ICU) (including intermediate care unit) with severe community-acquired pneumonia (CAP).

CAP is the sixth most common cause of death (acute mortality) in the United States and the leading cause of community-acquired infection requiring intensive care unit (ICU) admission. Despite significant advancements in medical care, there has been little change in crude mortality from respiratory tract infection for more than 5 decades (1950-2000). In the United States alone, over 1.3 million people were admitted to the hospital in 2002 with severe CAP (262 per 10,000 population) with an estimated inpatient cost of approximately $4.4 billion. In addition, severe CAP patients surviving hospitalization experience a significant increase in long-term morbidity (cardiovascular complications, impaired functional status, and recurrent hospitalizations) and a sizable mortality up to 1 year (up to 25%) that is independent of patient's chronic health condition.

Dysregulated systemic inflammation, characterized by persistent elevation in circulating inflammatory cytokine levels over time, is the central pathogenetic process contributing to short- and long-term morbidity and mortality in patients with severe CAP. Even when patients survive ICU and hospital admission, elevation in inflammatory cytokine lasts for greater than 3 weeks, and interleukin (IL)-6 levels at hospital discharge predict subsequent mortality. Endogenous and exogenous glucocorticoids are the most important physiologic inhibitors of inflammation. In a meta-analysis of four, small, published studies that included a total of 198 patients with severe CAP, prolonged glucocorticoid treatment was associated with a significant reduction in short-term mortality (RR = 0.40, 95%CI 0.18-0.89; p = 0.03; I2 12%). This Cooperative Studies Program (CSP) study will be the first large-scale, prospective, randomized clinical trial evaluating the efficacy of prolonged methylprednisolone in the treatment of severe CAP.

In this study, at each site, patients with severe CAP will be randomized in a 1:1 ratio to receive methylprednisolone or placebo in a double-blind fashion. The investigators have chosen a total duration of treatment of 20 days (7 days full dose followed by slow reduction over 13 days) to forestall relapse of systemic inflammation and allow recovery of the suppressed hypothalamic-pituitary-adrenal (HPA) axis. All patients will also receive standardized management of CAP in accordance with current practice guidelines. Randomization will be stratified separately within each participating site by whether or not the patient requires mechanical ventilation at the time of randomization. Patients will be followed clinically for 180 days. The primary outcome is all cause 60-day mortality. Secondary outcomes are (1) in-hospital morbidity-mortality, including ventilator-free days, multiorgan dysfunction syndrome (MODS)-free days, duration of ICU and hospital stay, and hospital discharge; and (2) posthospital discharge morbidity-mortality, including cardiovascular complications, functional and general health status in the first 180 days, rehospitalization, and mortality at 1 year. Serial blood samples will also be collected and stored for future translational research relating longitudinal inflammation markers to clinical outcomes.

Based on published studies and VA Decision Support System, the investigators estimate the all cause 60-day mortality in severe CAP patients admitted to ICU is 28%. The investigators hypothesize that prolonged methylprednisolone treatment will reduce the 60-day mortality from 28% to 21% (a 25% relative reduction). A total of 1406 patients (703 per group) will be required to give 85% power to detect this hypothesized improvement, using a two-sided 5% significance level test. Adjusting for 1% attrition, the target sample size is 1420. Assuming 5 years of accrual and an intake rate of 8 patients per year per Veterans Affairs Medical Center (VAMC), the investigators will need 36 participating VAMCs.

Treatment of severe CAP is of particular importance to the VA health care system because of the large patient population and because a single episode of severe CAP is associated with significant short- and long-term morbidity and mortality. In fiscal year 2006, 17,890 patients were admitted to the VA hospital system with a diagnosis of CAP. Of these, 3727 (21%) required ICU admission during their hospital stay. For ICU-admitted patients, mortality rates in the hospital at 60, 90, 180, and 365 days were 26%, 34%, 37%, 44%, and 51%, respectively. They had on average a hospital stay of 17.7 days with hospital costs of $49,936, and 48% of them were readmitted within 12 months of hospital discharge. This study will investigate the effects of an off-patent, inexpensive treatment that, based on strong experimental and translational evidence and the encouraging findings of preliminary trials, has the potential of significantly decreasing mortality and morbidity. Equally important, this study will advance knowledge on the relationship between inflammation and long-term outcome in severe CAP. Given that methylprednisolone is off-patent, there is little incentive for the pharmaceutical industry to fund this study. The VA system with its Cooperative Studies Program is uniquely suited to conduct the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient's origin. Patients are classified as having Community Acquired Pneumonia (CAP) if they are admitted directly from outside the hospital, including private residence, nursing home, rehabilitation center, other long-term care facility (health care-associated pneumonia (HCAP)).
* Clinical diagnosis of CAP.
* Have radiographically confirmed pneumonia (new or progressive pulmonary infiltrate(s) on chest radiograph or chest computed tomography scan consistent with bacterial pneumonia) AND have acute illness ( <=7 days' duration) with at least three of the following clinical signs or symptoms consistent with a lower respiratory tract infection:

New or increased cough Purulent sputum or change in sputum character Auscultatory findings consistent with pneumonia (e.g., rales, egophony, findings of consolidation) Dyspnea, tachypnea, or hypoxemia (O2 saturation <90% on room air or PaO2 <60 mmHg) Fever >= 38 C oral (>=38.5 C rectally or tympanically) or hypothermia (<=36 C) White blood cell count greater than 10,000 cells/mm3 or less than 4,000 cells/mm3 Greater than 15% immature neutrophils (bands) irrespective of WBC count

* Diagnosis of severe CAP. Pneumonia of sufficient severity to require admission to the ICU (including intermediate care unit) and meeting >=1 major or >= 3 minor modified Infectious Diseases Society of America (IDSA)/American

Thoracic Society (ATS) criteria.:

* 1 Major Criteria

  1. Use of invasive or noninvasive mechanical ventilation
  2. Vasopressors for shock despite adequate fluid resuscitation
  3. Arterial pH < 7.30 -OR >=3 Minor Criteria

  <!-- -->

  1. New onset of confusion or disorientation
  2. Hypothermia (core temperature <=36 C)
  3. Respiratory rate >=30 breaths/min
  4. Hypotension requiring aggressive fluid resuscitation
  5. Uremia (BUN >=20 mg/dL)
  6. PaO2: FiO2 ratio <=250 or SaO2:FiO2 ratio <=250
  7. Leukopenia (WBC count < 4000 cells/mm3)
  8. Platelet count < 100,000 cells/mm3 or > 400,000 cells/mm3
  9. Multilobar infiltrates

     Exclusion Criteria:

     - Patient's age 17 years or younger.

     - Vasopressor-dependent shock requiring moderate-to-high dose vasopressor (i.e., norepinephrine >=0.3 mcg/Kg/min) treatment for greater than 2 hours in patient that is adequately fluid-resuscitated (at least 4 liters of crystalloids) WITH central venous pressure (CVP) equal to or greater than 8 mm Hg for nonventilated patients and equal to or greater than 12 mm Hg for ventilated patients. (See explanation below)*

     - Major gastrointestinal bleeding requiring transfusion of 5 units or more of packed red blood cells within 3 months of current hospitalization.

     - Any condition requiring 20 mg of prednisone equivalent/day for greater than 14 days, over the last 3 months.

     - Chronic obstructive pulmonary disease (COPD) with acute exacerbation requiring glucocorticoid treatment at hospital admission. Patients with short-term glucocorticoid use (e.g., methylprednisolone up to 300 mg within 5 days of randomization) will not be excluded.

     - Patients enrolled in another experimental (interventional) protocol.

     - Pregnancy, confirmed by urine or serum test.

     - Presence of postobstructive pneumonia or cystic fibrosis.

     - Clinical history consistent with aspiration of gastric content (i.e., loss of consciousness or seizure).

     - Active tuberculosis or fungal infection.

     - Moribund patient (i.e., not expected to live more than 24 h) or with recent (within 7 days) cardiopulmonary arrest, or with (known or suspected) irreversible cessation of all brain function, or comfort measure status.

     - Presence of preexisting medical condition that is irreversible and expected to be fatal within 3 months.
     * Patients with severe immunosuppression (i.e., HIV with CD4 <200), neutropenia (less than 1000 neutrophils) not related to pneumonia, acute burn injury, or receiving immunosuppressive or cytotoxic therapy for any reason.
     * Chronic severe cognitive impairment caused by dementia or central nervous system pathologies (tumor, cerebro-vascular accident, infections, or head injuries) as defined by the site investigator by obtaining medical history and reviewing medical record.
     * The physician doesn't feel the patient is a viable candidate for the study (e.g., presence of hypersensitivity or previous severe adverse reaction to cosyntropin or any glucocorticoid, history of adrenal insufficiency or chronic systemic steroid use placing the patient at risk for relative adrenal insufficiency).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco U Meduri, MD, Study Chair — Memphis VA Medical Center, Memphis, TN
Locations (30):
- United States (29):
  - Phoenix VA Health Care System Carl T. Hayden VA Medical Center, Phoenix, AZ, Phoenix, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Robley Rex VA Medical Center, Louisville, KY, Louisville, Kentucky
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - VA Sierra Nevada Health Care System, Reno, NV, Reno, Nevada
  - VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Oklahoma City VA Medical Center, Oklahoma City, OK, Oklahoma City, Oklahoma
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia SC, Columbia, South Carolina
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meduri GU, Shih MC, Bridges L, Martin TJ, El-Solh A, Seam N, Davis-Karim A, Umberger R, Anzueto A, Sriram P, Lan C, Restrepo MI, Guardiola JJ, Buck T, Johnson DP, Suffredini A, Bell WA, Lin J, Zhao L, Uyeda L, Nielsen L, Huang GD; ESCAPe Study Group. Low-dose methylprednisolone treatment in critically ill patients with severe community-acquired pneumonia. Intensive Care Med. 2022 Aug;48(8):1009-1023. doi: 10.1007/s00134-022-06684-3. Epub 2022 May 13. PMID 35723686

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Inactive Substance | Arm 2: Methylprednisolone
Started | 287 | 297
Completed | 169 | 180
Not Completed | 118 | 117
Not completed — Death | 83 | 78
Not completed — Study ended early | 23 | 26
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Patient Withdrawn by LAR/DPOA | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Inactive Substance: Inactive substance
  Inactive substance will be given in a double-blind fashion for 20 full days. The treatment course includes a bolus dose on the day of randomization, 7 days of full dose (40 mg/day), 7 days of half dose (20 mg/day), and 6 days of tapering doses (12 mg/day and 4 mg/day).
- Total: Total of all reporting groups
Arm/Group | Arm 1: Inactive Substance | Arm 2: Methylprednisolone | Total
Number analyzed (Participants) | 287 | 297 | 584
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant in Arm 1 was missing the demographic information form.
  years
    number analyzed (Participants) | 286 | 297 | 583
    (all) | 68.6 (11.1) | 69.0 (10.8) | 68.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in Arm 1 was missing the demographic information form.
  Participants
    number analyzed (Participants) | 286 | 297 | 583
    Female | 13 | 8 | 21
    Male | 273 | 289 | 562
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Eleven participants in Arm 1, and six participants in Arm 2 were missing information on ethnicity.
  Participants
    Ethnicity: number analyzed (Participants) | 280 | 286 | 566
    Ethnicity: Not Spanish, Hispanic or Latino | 251 | 255 | 506
    Ethnicity: Mexican, Mexican American, or Chicano | 12 | 16 | 28
    Ethnicity: Puerto Rican | 8 | 5 | 13
    Ethnicity: Cuban | 1 | 0 | 1
    Ethnicity: Other Spanish, Hispanic, or Latino | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race is check all that apply. Therefore, the numbers for individual categories do not add up to the number of patient randomized.
  Participants
    White: number analyzed (Participants) | 281 | 287 | 568
    White | 227 | 245 | 472
    Black/African American: number analyzed (Participants) | 281 | 287 | 568
    Black/African American | 48 | 36 | 84
    Other: number analyzed (Participants) | 281 | 287 | 568
    Other | 10 | 15 | 25
BMI >=30 [Count of Participants; unit: Participants] — Population: Two participants in Arm 1 are missing this value.
  Participants
    number analyzed (Participants) | 285 | 297 | 582
    Yes | 70 | 62 | 132
    No | 215 | 235 | 450
Mechanical Ventilation at Study Entry [Count of Participants; unit: Participants]
  Yes | 96 | 97 | 193
  No | 191 | 200 | 391
SOFA Score [Mean (Standard Deviation); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) is a morbidity severity score and mortality estimation tool developed from a large sample of ICU patients throughout the world. The "worst" measurement was defined as the measure that correlated to the highest number of points. The SOFA score ranges from 0 to 24. Population: The number analyzed in Arm 1 is different from the overall due to missing values.
  units on a scale
    number analyzed (Participants) | 285 | 297 | 582
    (all) | 6.29 (2.85) | 6.68 (3.0) | 6.49 (2.93)
Vasopressor Dependent Shock at or Prior to Study Entry [Count of Participants; unit: Participants] — Population: The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 285 | 296 | 581
    Yes | 32 | 44 | 76
    No | 253 | 252 | 505
Any Major Co-Morbidities [Count of Participants; unit: Participants] — Population: The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 285 | 297 | 582
    Yes | 275 | 290 | 565
    No | 10 | 7 | 17
Number of Major Co-Morbidities [Mean (Standard Deviation); unit: Comorbidities] — The range for number of co-morbidities was 0-9, with 9 being the highest number of comorbidities. Population: The number analyzed is different from the overall due to missing values.
  Comorbidities
    number analyzed (Participants) | 285 | 297 | 582
    (all) | 3.9 (1.9) | 4.0 (1.8) | 4.0 (1.8)
Charlson Comorbidity Index [Mean (Standard Deviation); unit: comorbidity score] — The Charleston Comorbidity Index identifies 17 comorbidities that are associated with mortality and appropriately assigns weights to each of them, ranging from 1 to 6 points. The final score is obtained via the summation of applicable points and ranges from 0 (no disease burden) to 29 (maximal disease burden). Population: The number analyzed is different from the overall due to missing values.
  comorbidity score
    number analyzed (Participants) | 285 | 297 | 582
    (all) | 5.65 (2.24) | 5.77 (2.39) | 5.71 (2.32)
ACE 27 Overall Comorbidity Score [Count of Participants; unit: Participants] — Population: The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 285 | 297 | 582
    0 (None) | 8 | 6 | 14
    1 (Mild) | 33 | 38 | 71
    2 (Moderate) | 59 | 51 | 110
    3 (Severe) | 185 | 202 | 387
ACE 27 total score [Mean (Full Range); unit: units on a scale] — The overall ACE-27 score also ranges from none (0) to severe (3). Population: The number analyzed is different from the overall due to missing values.
  units on a scale
    number analyzed (Participants) | 285 | 297 | 582
    (all) | 2.48 [0 to 3] | 2.51 [0 to 3] | 2.50 [0 to 3]
Karnofsky Performance Score [Mean (Full Range); unit: units on a scale] — The Karnofsky Performance Score (KPS) ranking runs from 100 to 0, where 100 is "perfect" health and 0 is death. Population: The number analyzed is different from the overall due to missing values.
  units on a scale
    number analyzed (Participants) | 280 | 291 | 571
    (all) | 72.9 [20 to 100] | 72.4 [20 to 100] | 72.6 [20 to 100]
Health Care Associated Pneumonia [Count of Participants; unit: Participants]
  Pts. w/No HCAP (%) | 198 | 185 | 383
  Pts. with HCAP (%) | 89 | 112 | 201
Admission from the Ward [Count of Participants; unit: Participants]
  Pts. Admitted from Ward (%) | 57 | 66 | 123
  Pts. not Admitted from Ward (%) | 230 | 231 | 461
Pneumonia Severity Index (PSI) Score [Mean (Standard Deviation); unit: Severity Score] — The purpose of the Pneumonia Severity Index (PSI) Score is to classify the severity of a patient's pneumonia. Scores range from 0 to >130. For scores over 90, hospitalization may be recommended/necessary. Population: The number analyzed is different from the overall due to missing values.
  Severity Score
    number analyzed (Participants) | 286 | 297 | 583
    (all) | 122.3 (34.4) | 125.6 (37.2) | 124.0 (35.8)
Pneumonia Severity Index (PSI) Class [Count of Participants; unit: Participants] — The purpose of the Pneumonia Severity Index (PSI) Score is to classify the severity of a patient's pneumonia. The Risk Class ranges from Class I (Low Risk) to Class V (High Risk). Population: Risk Class I to Risk Class III indicate lower risk; Risk Class IV to V require hospitalization.
  The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 285 | 297 | 582
    I | 4 | 3 | 7
    II | 13 | 13 | 26
    III | 29 | 41 | 70
    IV | 126 | 121 | 247
    V | 113 | 119 | 232
Chest Radiographic Score [Mean (Full Range); unit: units on a scale] — The range for Alveolar Consolidation is 0 to 4, where 0 is no Alveolar Consolidation, up to Alveolar Consolidation in 4 quadrants. Population: The number analyzed is different from the overall due to missing values.
  units on a scale
    number analyzed (Participants) | 282 | 294 | 576
    (all) | 1.94 [0 to 4] | 2.09 [0 to 4] | 2.02 [0 to 4]
Chest Radiograph Class [Count of Participants; unit: Participants] — Population: The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 282 | 294 | 576
    No Alveolar Consolidation | 15 | 13 | 28
    Alveolar Consolidation, 1 quadrant | 93 | 68 | 161
    Alveolar Consolidation, 2 quadrants | 103 | 127 | 230
    Alveolar Consolidation, 3 quadrants | 36 | 52 | 88
    Alveolar Consolidation, 4 quadrants | 35 | 34 | 69
Bilateral Involvement [Count of Participants; unit: Participants] — Population: The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 276 | 288 | 564
    Bilateral Involvement | 163 | 189 | 352
    No Bilateral Involvement | 113 | 99 | 212
PaO2:FiO2 (If PaOD is available) [Mean (Standard Deviation); unit: mmHg] — PaO2/FiO2 ratio is the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage). Lower scores are more severe, and show a higher risk for mortality. Population: The number analyzed is different from the overall due to missing values.
  mmHg
    number analyzed (Participants) | 178 | 201 | 379
    (all) | 188 (90) | 181 (85) | 184 (87)
SpO2:FiO2 (if PaO2 is not available) [Mean (Standard Deviation); unit: mmHg] — When the PaO2 is unknown because an Arterial Blood Gas (ABG) test is not available, the SpO2 measured by pulse oximetry can be used to approximate the PaO2. Population: The number analyzed is different from the overall due to missing values.
  mmHg
    number analyzed (Participants) | 88 | 79 | 167
    (all) | 286 (98) | 283 (101) | 284 (99)
ALI/ARDS at randomization [Count of Participants; unit: Participants] — Population: The number analyzed is different from the overall due to missing values.
  Participants
    number analyzed (Participants) | 285 | 297 | 582
    Yes | 39 | 26 | 65
    No | 246 | 271 | 517

OUTCOME MEASURES:

1. Primary Outcome: 60-day Mortality
Description: The primary outcome is all-cause mortality at 60 days, defined by whether the patient has died by the end of study day 60.
Time Frame: 60-day
Population: Numbers provided are overall and by stratum.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Inactive Substance | Arm 2: Methylprednisolone
Number analyzed (Participants) | 287 | 297
Participants
  Died on or prior to study day 60: Yes | 50 | 47
  Died on or prior to study day 60: No | 227 | 239
  Died on or prior to study day 60: Unknown | 10 | 11
  On Mechanical Ventilation at Study Entry: number analyzed (Participants) | 96 | 97
  On Mechanical Ventilation at Study Entry: Yes | 24 | 22
  On Mechanical Ventilation at Study Entry: No | 70 | 72
  On Mechanical Ventilation at Study Entry: Unknown | 2 | 3
  Not on Mechanical Ventilation: number analyzed (Participants) | 191 | 200
  Not on Mechanical Ventilation: Yes | 26 | 25
  Not on Mechanical Ventilation: No | 157 | 167
  Not on Mechanical Ventilation: Unknown | 8 | 8
Statistical Analysis 1: Comparison: Arm 1: Inactive Substance vs Arm 2: Methylprednisolone; Test type: Superiority; p = 0.635, Mantel Haenszel; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.58 to 1.40]

ADVERSE EVENTS:
Time Frame: All SAEs were reported from Randomization to day 180.
Description: We did not collect data on non-serious adverse events.
Groups:
- Arm 1: Inactive Substance: Inactive substance
  Methylprednisolone: Methylprednisolone will be given in a double-blind fashion for 20 full days. The treatment course includes a bolus dose on the day of randomization, 7 days of full dose (40 mg/day), 7 days of half dose (20 mg/day), and 6 days of tapering doses (12 mg/day and 4 mg/day).
Arm/Group | Arm 1: Inactive Substance | Arm 2: Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 84/287 | 79/297
Serious Adverse Events (participants affected / at risk) | 162/287 | 167/297
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Inactive Substance (N=287) | Arm 2: Methylprednisolone (N=297)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Blood disorder (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 6 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 4
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 5 | 1
Cardiac failure congestive (Cardiac disorders) | 18 | 25
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Chordae tendinae rupture (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 0 | 1
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 3
Complication associated with device (General disorders) | 0 | 1
Death (General disorders) | 1 | 2
Impaired healing (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 5 | 9
Non-cardiac chest pain (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 2 | 0
Vascular stent restenosis (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatitis chronic active (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 3 | 4
Clostridium difficile infection (Infections and infestations) | 0 | 2
Clostridium difficile sepsis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 1
Gangrene (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Meningitis listeria (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pancreatic abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 38 | 27
Pneumonia bacterial (Infections and infestations) | 1 | 1
Pneumonia cryptococcal (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 2
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 4
Septic shock (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 6
Urosepsis (Infections and infestations) | 0 | 1
Vaccine breakthrough infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Laboratory test abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Basal ganglia stroke (Nervous system disorders) | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 6
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 2
Myoclonic epilepsy (Nervous system disorders) | 0 | 1
Myxoedema coma (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 2 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Vascular dementia (Nervous system disorders) | 1 | 0
Unintentional medical device removal (Product Issues) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 3 | 4
Delirium tremens (Psychiatric disorders) | 1 | 1
Drug abuse (Psychiatric disorders) | 0 | 1
Drug dependence (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 4 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 6 | 11
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 3
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Pulmonary renal syndrome (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Medical device battery replacement (Surgical and medical procedures) | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 2
Withdrawal of life support (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Dry gangrene (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 3
Shock (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes